CLINICAL TRIAL: NCT06311383
Title: A Non-interventional Study for Women With HR-positive, HER2-negative Locally Advanced or Metastatic Breast Cancer to Evaluate the Real-world Effectiveness of Treatment Algorithms Beginning With Kisqali (Ribociclib) in Combination With an Aromatase Inhibitor/Fulvestrant, or With Endocrine Therapy or Chemotherapy as First Line Treatment
Brief Title: A Non-interventional Study for Women With HR-positive, HER2-negative Locally Advanced or Metastatic Breast Cancer to Evaluate the Real-world Effectiveness of Treatment Algorithms Beginning With Ribociclib + AI/FUL, or With Endocrine Therapy or Chemotherapy as First Line Treatment
Acronym: RIBANNA
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011ADE03
Record Dates: First submitted 2023-12-29; First posted 2024-03-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; NIS; Ribociclib; Metastatic Breast Cancer; HR+; HER2-; Real World Evidence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- First-line Ribociclib + endocrine therapy: Ribociclib + letrozole, or Ribociclib + anastrozole, or Ribociclib + exemestane, or Ribociclib + fulvestrant
  Interventions: Drug: First-line Ribociclib + endocrine therapy
- First-line endocrine therapy: As of physicians choice
  Interventions: Drug: First-line endocrine therapy
- First-line chemotherapy: As of physicians choice
  Interventions: Drug: First-line chemtherapy

INTERVENTIONS:
Drug: First-line Ribociclib + endocrine therapy — Ribociclib + letrozole, or Ribociclib + anastrazole, or Ribociclib + exemestane, or Ribociclib + fulvestrant
  Groups: First-line Ribociclib + endocrine therapy
Drug: First-line endocrine therapy — As of physicians choice
  Groups: First-line endocrine therapy
Drug: First-line chemtherapy — As of physicians choice
  Groups: First-line chemotherapy

SUMMARY:
This is a non-interventional observational study conducted in Germany to evaluate the real-world effectiveness, tolerability, safety, and quality of life in patients with locally advanced/metastatic HR+/HER2- breast cancer treated with one of the following 1st line treatments: Ribociclib + AI/FUL, or endocrine monotherapy, or chemotherapy

DETAILED DESCRIPTION:
This non-interventional study collects data from clinical practice capturing on effectiveness, safety and tolerability, duration of therapy, and quality of life of ribociclib in combination with an aromatase inhibitor/fulvestrant in daily routine and in line with the respective current German summary of product characteristics. In order to put these results into perspective, data is also collected on patients treated with endocrine therapy or chemotherapy for first line locally advanced or metastatic breast cancer. To gain insight into algorithms and outcome of sequential therapy, up to three lines of treatment are documented within this study. The information gathered and evaluated in this NIS is helping to answer open questions for the treatment of locally advanced/metastatic breast cancer and provides first insights into the treatment reality with ribociclib in this setting. This includes, but is not limited to, the questions on baseline demographics leading to a specific treatment decision, as well as efficacy and clinical routine related to treatment sequencing. In addition, data on the mutation status (including PIK3CA and BRCA1/2) is collected at different time points to generate insights into the clinical routine of mutation testing and to understand its impact on therapy sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histological diagnosis of locally advanced/metastatic HR+/HER2- breast cancer. Histological diagnosis does not necessarily origin from metastasis, but must reflect the most recent disease status
* No prior systemic treatment for locally advanced/metastatic disease in the palliative setting
* The treating physician has made the decision to treat the patient
* with ribociclib in combination with an aromatase inhibitor or fulvestrant as initial treatment in first line, or
* endocrine therapy as initial treatment in first line (e.g. letrozole, anastrozole, fulvestrant), or
* chemotherapy as initial treatment in first line (e.g. taxanes, capecitabine, with or without bevacizumab)
* Written informed consent of the patient
* Patient who initiated treatment for first line no longer than 4 weeks (28 days) prior to written informed consent for this study
* Planned treatment is in line with the respective current German SmPC ("Summary of product characteristics")
* Patient is ≥18 years

Exclusion Criteria:

* Patients unable to provide written informed consent
* Contra-indication according to the respective current German SmPC ("Summary of product characteristics"), as judged by the treating physician
* The patient is currently under active treatment in an investigational study

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult females with HR+/HER2- locally advanced/metastatic breast cancer (progressed following prior therapy or de novo). Hereby locally advanced is defined by the following criteria (at least one must apply): tumor size > 5 cm (T3), skin or chest wall infiltration (T4a, T4b), inflammatory breast cancer (T4c), fixed axilla-located lymph node conglomerate or intraclavicular lymph node metastasis (cN3; German S3 guideline for early detection, diagnosis, therapy and follow-up care of breast cancer; Version 4.1.2018). Patients are classified as therapy naïve for locally advanced/metastatic disease if they have not yet received a systemic therapy in the palliative setting. Patients with locally advanced breast cancer who have received therapy-(lines) in the adjuvant/curative setting are eligible after progression to e.g. a metastatic breast cancer. All patients who already received a palliative therapy for locally advanced/metastatic breast cancer are excluded from study participation.
Sampling Method: Non-Probability Sample
Enrollment: 2610 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 88 months
  Progression-free survival was defined as first intake of study medication in current-line therapy up to first documented progress or death from any cause in this treatment line. If a patient had not had an event, progression-free survival was censored at the end of the respective therapy line.

SECONDARY OUTCOMES:
Sequential progression-free survival (PFS_S) | Up to 88 months
  Sequential progression-free survival up to second-line therapy was defined as time between first intake of study medication in first-line therapy up to progress or death after second-line therapy. Sequential progression-free survival up to third-line therapy was defined as time between first intake of study medication in first-line therapy up to progress or death after third-line therapy. Sequential progression-free survival for all further therapy lines were analyzed according to the definitions above.
Time to treatment failure (TTF) | Up to 88 months
  Time to treatment failure (TTF) from current-line therapy was defined as time between first intake of study medication in current-line therapy up to therapy discontinuation because of progress, adverse events leading to discontinuation or death.
Time to first chemotherapy | Up to 88 months
  Time to first chemotherapy was defined as time between first intake of study medication in first-line therapy up to first application of chemotherapy for patients enrolled in 1st line option ribociclib + AI/FU or endocrine therapy.
Time to next treatment / therapy (TTNT) after 1st line treatment | Up to 88 months
  Time to next treatment / therapy (TTNT) was defined as time between first intake of study medication in first-line therapy up to first intake of medication in the next therapy line.
Overall survival (OS) | Up to 88 months
  Overall survival (OS) was defined as time between first intake of study medication in first-line therapy up to death from any cause. If a patient was not known to have died, survival was censored at the date of last contact.
Dose reduction | Up to 88 months
  Dose reduction rates and reasons
Dose interruption | Up to 88 months
  Dose interruption rates and reasons
Discontinuations | Up to 88 months
  Discontinuations rates and reasons
Adherence - MMAS-8 questionnaire | Up to 87 weeks
  Patient adherence for ribociclib was assessed using the MMAS-8 questionnaire. This questionnaire was only send to patients enrolled in the first-line option ribociclib + AI/FU. The score was analyzed using descriptive statistics and adherence categories low, medium and high were displayed by visit. Questionnaires were only included if all questionnaire items were answered.
  The total scale has a range of 0 to 8.0 where:
  * Low Adherence (< 6)
  * Medium Adherence (6 to <8)
  * High Adherence (= 8)
Number of participants with mutations | Up to 88 months
  Number of participants with mutations will be collected
Quality of life for specific cohorts and treatment lines - EORTC QLQ-C30 | Up to 88 months
  Quality of life during documented therapy lines was assessed using the EORTC QLQ-C30. Scale and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life for specific cohorts and treatment lines - EORTC QLQ-BR23 | Up to 88 months
  Quality of life during documented therapy lines was assessed using the EORTC QLQ-BR23. Scale and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life for specific cohorts and treatment lines - HADS-D | Up to 88 months
  Quality of life during documented therapy lines was assessed using the HADS-D. Scale ranges between 0 and 21, a high score means a high level of anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (224):
- Germany (224):
  - Novartis Investigative Site, Baden-Baden, Baden-Wurttemberg
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Freudenstadt, Baden-Wurttemberg
  - Novartis Investigative Site, Heidenheim, Baden-Wurttemberg
  - Novartis Investigative Site, Karlsruhe, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Mutlangen, Baden-Wurttemberg
  - Novartis Investigative Site, Nürtingen, Baden-Wurttemberg
  - Novartis Investigative Site, Ostfildern, Baden-Wurttemberg
  - Novartis Investigative Site, Pforzheim, Baden-Wurttemberg
  - Novartis Investigative Site, Reutlingen, Baden-Wurttemberg
  - Novartis Investigative Site, Rottweil, Baden-Wurttemberg
  - Novartis Investigative Site, Schwäbisch Hall, Baden-Wurttemberg
  - Novartis Investigative Site, Sigmaringen, Baden-Wurttemberg
  - Novartis Investigative Site, Winnenden, Baden-Wurttemberg
  - Novartis Investigative Site, Altötting, Bavaria
  - Novartis Investigative Site, Amberg, Bavaria
  - Novartis Investigative Site, Ansbach, Bavaria
  - Novartis Investigative Site, Aschaffenburg, Bavaria
  - Novartis Investigative Site, Augsburg, Bavaria
  - Novartis Investigative Site, Bamberg, Bavaria
  - Novartis Investigative Site, Bayreuth, Bavaria
  - Novartis Investigative Site, Donauwörth, Bavaria
  - Novartis Investigative Site, Ebersberg, Bavaria
  - Novartis Investigative Site, Eggenfelden, Bavaria
  - Novartis Investigative Site, Kempten (Allgäu), Bavaria
  - Novartis Investigative Site, Kronach, Bavaria
  - Novartis Investigative Site, Krumbach, Bavaria
  - Novartis Investigative Site, Landshut, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Nuremberg, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Straubing, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Mannheim, Beden Wuerttenberg
  - Novartis Investigative Site, Brandenburg, Brandenburg
  - Novartis Investigative Site, Cottbus, Brandenburg
  - Novartis Investigative Site, Doberlug-Kirchhain, Brandenburg
  - Novartis Investigative Site, Fürstenwalde, Brandenburg
  - Novartis Investigative Site, Ludwigsfelde, Brandenburg
  - Novartis Investigative Site, Spremberg, Brandenburg
  - Novartis Investigative Site, Bremen, City state Bremen
  - Novartis Investigative Site, Bremerhaven, City state Bremen
  - Novartis Investigative Site, Schwerte, Germany
  - Novartis Investigative Site, Wiesbaden, Germany
  - Novartis Investigative Site, Hamburg, Hamburg
  - Novartis Investigative Site, Bad Homburg, Hesse
  - Novartis Investigative Site, Bad Nauheim, Hesse
  - Novartis Investigative Site, Darmstadt, Hesse
  - Novartis Investigative Site, Erbach im Odenwald, Hesse
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Langen, Hesse
  - Novartis Investigative Site, Lich, Hesse
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Braunschweig, Lower Saxony
  - Novartis Investigative Site, Buchholz, Lower Saxony
  - Novartis Investigative Site, Damme, Lower Saxony
  - Novartis Investigative Site, Georgsmarienhütte, Lower Saxony
  - Novartis Investigative Site, Hamelin, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Hildesheim, Lower Saxony
  - Novartis Investigative Site, Ilsede, Lower Saxony
  - Novartis Investigative Site, Lingen Ems, Lower Saxony
  - Novartis Investigative Site, Osnabrück, Lower Saxony
  - Novartis Investigative Site, Rotenburg (Wümme), Lower Saxony
  - Novartis Investigative Site, Twistringen, Lower Saxony
  - Novartis Investigative Site, Westerstede, Lower Saxony
  - Novartis Investigative Site, Wolfenbüttel, Lower Saxony
  - Novartis Investigative Site, Neubrandenburg, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Rostock, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Schwerin, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Stralsund, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Arnsberg, North Rhine-Westphalia
  - Novartis Investigative Site, Bergisch Gladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Bielefeld, North Rhine-Westphalia
  - Novartis Investigative Site, Bochum, North Rhine-Westphalia
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dortmund, North Rhine-Westphalia
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Gelsenkirchen, North Rhine-Westphalia
  - Novartis Investigative Site, Hagen, North Rhine-Westphalia
  - Novartis Investigative Site, Herdecke, North Rhine-Westphalia
  - Novartis Investigative Site, Herne, North Rhine-Westphalia
  - Novartis Investigative Site, Hilden, North Rhine-Westphalia
  - Novartis Investigative Site, Krefeld, North Rhine-Westphalia
  - Novartis Investigative Site, Lemgo, North Rhine-Westphalia
  - Novartis Investigative Site, Mönchengladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Olpe, North Rhine-Westphalia
  - Novartis Investigative Site, Paderborn, North Rhine-Westphalia
  - Novartis Investigative Site, Remscheid, North Rhine-Westphalia
  - Novartis Investigative Site, Siegen, North Rhine-Westphalia
  - Novartis Investigative Site, Troisdorf, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Wesel, North Rhine-Westphalia
  - Novartis Investigative Site, Witten, North Rhine-Westphalia
  - Novartis Investigative Site, Mayen, Rhineland-Palatinate
  - Novartis Investigative Site, Neustadt an der Weinstraße, Rhineland-Palatinate
  - Novartis Investigative Site, Simmern, Rhineland-Palatinate
  - Novartis Investigative Site, Lebach, Saarland
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Lohsa-Weisskollm, Saxony
  - Novartis Investigative Site, Neustadt in Sachsen, Saxony
  - Novartis Investigative Site, Pirna, Saxony
  - Novartis Investigative Site, Plauen, Saxony
  - Novartis Investigative Site, Rodewisch, Saxony
  - Novartis Investigative Site, Scheibenberg, Saxony
  - Novartis Investigative Site, Schkeuditz, Saxony
  - Novartis Investigative Site, Zittau, Saxony
  - Novartis Investigative Site, Zxickau, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
  - Novartis Investigative Site, Quedlinburg, Saxony-Anhalt
  - Novartis Investigative Site, Flensburg, Schleswig-Holstein
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Berlin, State of Berlin
  - Novartis Investigative Site, Apolda, Thuringia
  - Novartis Investigative Site, Eisenach, Thuringia
  - Novartis Investigative Site, Erfurt, Thuringia
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Meiningen, Thuringia
  - Novartis Investigative Site, Mühlhausen, Thuringia
  - Novartis Investigative Site, Nordhausen, Thuringia
  - Novartis Investigative Site, Suhl, Thuringia
  - Novartis Investigative Site, Altötting
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Liebenwerda
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Brandenburg
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Bremerhaven
  - Novartis Investigative Site, Celle
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Eutin
  - Novartis Investigative Site, Friedberg
  - Novartis Investigative Site, Friedrichshafen
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Goch
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Gummersbach
  - Novartis Investigative Site, Halberstadt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hamelin
  - Novartis Investigative Site, Hanau
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Hof
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Kulmbach
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Loerrach
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Marktredwitz
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Naunhof
  - Novartis Investigative Site, Neuruppin
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Passau
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rheine
  - Novartis Investigative Site, Rodgau
  - Novartis Investigative Site, Rosenheim
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Saarlouis
  - Novartis Investigative Site, Salzgitter
  - Novartis Investigative Site, Schkeuditz
  - Novartis Investigative Site, Schorndorf
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Schweinfurt
  - Novartis Investigative Site, Soest
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stendal
  - Novartis Investigative Site, Stolberg
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Suhl
  - Novartis Investigative Site, Torgau
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Vechta
  - Novartis Investigative Site, Völklingen
  - Novartis Investigative Site, Weiden
  - Novartis Investigative Site, Weinheim
  - Novartis Investigative Site, Wetzlar
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Wilhelmshaven
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Worms
  - Novartis Investigative Site, Würselen
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Decker T, Brucker C, Engel A, Fasching PA, Gohler T, Jackisch C, Janssen J, Kohler A, Ludtke-Heckenkamp K, Luftner D, Marme F, van Mackelenbergh M, Rautenberg B, Schmidt M, Weide R, Wimberger P, Kisseleff E, Pfister C, Roos C, Wilhelm N, Wockel A. Conditional progression-free survival in patients with metastatic hormone receptor-positive, human epidermal growth factor receptor 2-negative breast cancer treated with first-line ribociclib and endocrine therapy: real-world data from the RIBANNA study. ESMO Open. 2025 Jun;10(6):105105. doi: 10.1016/j.esmoop.2025.105105. Epub 2025 May 16. PMID 40381382